CLINICAL TRIAL: NCT05404035
Title: "Family Connections" an Intervention for Caregivers of People With Eating Disorders and Personality Disorders: Study Protocol for a Randomized Controlled Trial.
Brief Title: "Family Connections" for Caregivers of People With Eating Disorders and Personality Disorders.
Acronym: FC-ED&PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UV-1955599
Record Dates: First submitted 2022-05-23; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Relatives
Keywords: Intervention; family members; caregivers; eating disorders; personality disorders
MeSH Terms: conditions — Feeding and Eating Disorders; Personality Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial, Efficacy Study
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Connections for relatives of people with eating disorders and personality disorders (Experimental): The intervention lasts 3 months and includes 14 two-hour sessions with a group format on a weekly basis. The FC program is divided into 7 modules: 2 of Psychoeducation (ED and PD criteria, explanatory theories, available treatments, comorbidity with PD, etc.) and 5 modules of Dialectical Behavioral Therapy skills training (Relationship mindfulness, effective communication, aceptation, validation, problem management and meaning of life).
  Interventions: Behavioral: Family Connections for relatives of people with eating disorders and personality disorders
- Optimized Treatment As Usual (Active Comparator): Family members with this condition will continue to receive the usual treatment provided by their referral care center. In addition, we will optimize the treatment, with 3 two-hour psychoeducation sessions in group format each week (ED and PD, explanatory theories, available treatments, comorbidity with PD).
  Interventions: Behavioral: Optimized Treatment As Usual

INTERVENTIONS:
Behavioral: Family Connections for relatives of people with eating disorders and personality disorders — The FC program (Fruzzetti and Hoffman, 2005) is divided into 7 modules:
  1. Introduction to the intervention program. Program objectives, guidelines, criteria, and symptoms of ED and PD.
  2. Psychoeducation on the development of ED and PD, explanatory theories, available treatments, comorbidity with PD.
  3. Emotional regulation skills and awareness, and to decrease emotional reactivity.
  4. Skills to improve the quality of relationships in family interactions (letting go of guilt and anger, acceptance skills in relationships).
  5. Communication skills and effective self-expression, such as validation.
  6. Problem management and making safe plans for crisis management.
  7. Making new sense of my relationship with my family member, an opportunity to grow together.
  All the modules include practice exercises, video viewing, and homework assignment.
  Arms: Family Connections for relatives of people with eating disorders and personality disorders
Behavioral: Optimized Treatment As Usual — Family members with this condition will continue to receive the usual treatment provided by their referral care center. In addition, we will optimize the treatment, following the recommendations of the international guidelines for the treatment of ED (NICE, 2017). There will be 3 two-hour session in group format each week, with the following components: Up-to-date information and research on ED and PD; Psychoeducation on the development of ED and PD; Explanatory theories; Available treatments and comorbidity.
  In both conditions, after each face-to-face session, the participant will be asked to review the contents addressed during the session as homework (independently of the homework corresponding to the specific module being addressed). All interventions carried out with family members will be performed by clinical psychologists or general health psychologists with at least a master's degree or a doctoral degree and previous training in the application of the programs.
  Arms: Optimized Treatment As Usual

SUMMARY:
The aim of our study is to verify the efficacy of the Family Connections intervention for relatives of people diagnosed with eating disorders and personality disorders in a randomized control trial with a Spanish participants.

DETAILED DESCRIPTION:
Eating disorders (EDs) are serious mental health problems that cause disturbances related to food intake and lead to major concerns about weight and body shape. In addition, they have an impact on social functioning and lead to psychological symptoms such as depression and anxiety, social isolation, interpersonal difficulties, low self-esteem, and reduced autonomy. These disorders share a high comorbidity with personality disorders (PD) that ranges from 27-93%, leading to increased severity and worse quality of life. Families of people with ED perceive a high burden of the illness and report mental health problems. Existing intervention programs specifically targeting caregivers of people with ED are based on psychoeducation, systemic cognitive-behavioral therapy, although specific treatments for family members of people with ED and PD are still scarce. However, a skills training program called "Family Connections" (FC) was developed by Hoffman and Fruzzetti's group for borderline personality disorder (BPD). It is a program consisting of 12 two-hour sessions that take place weekly. It is divided into six modules that include psychoeducation about the disorder and how it affects family functioning, and skills adapted from Dialectical Behavior Therapy, such as mindfulness, emotional regulation, validation, radical acceptance, and problem management, among others. In addition, all the modules include specific practical exercises, video examples, and homework. There is also a forum where family members build an emotional support network. So far, the results of this program in non-randomized clinical trials show significant decreases in the subjective experience of burden of illness, perceived distress, and depression, as well as improvements in coping strategies. The aims of this study are the following: (a) to adapt and test, in the Spanish population, the modules of the FC intervention protocol, designed to be applied specifically to relatives of patients with ED and PD; (b) to test the efficacy of FC in reducing the perceived burden of illness and clinical symptomatology in relatives of patients with ED and PD and improving family relationships and quality of life; (c) to test its efficiency, understood as the acceptance of the intervention program by the participants and clinicians, and demonstrate its viability; (d) to carry out an effective dissemination of this protocol. This paper presents the study protocol. The study design consists of a two-arm randomized controlled trial with two conditions: Family Connections (FC-ED & PD) or Treatment as usual optimized (TAU-O). Participants will be family members of patients with eating disorders and personality disorders (or dysfunctional personality traits) according to the 5th version of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). The caregivers' primary outcome measures will be the BAS and a Family-Patient Critical Incident Record. Secondary outcomes will be the EDSIS, FAD-GD, MEMs, MQLI, DASS-21, DERS, and QoL. The patients' primary outcome measures will be a Family-Patient Critical Incident Record, the EAT-26, PHQ-9, OASIS, VIRS, and LEAP. Participants will be assessed at pre-treatment, post-treatment, and twelve months follow-up. The intention-to-treat principle will be used when analyzing data, using mixed-effects models with full information and maximum likelihood estimation.

ELIGIBILITY:
Inclusion Criteria:

* Having a family member diagnosed with eating disorders and personality disorders (or personality disorder traits).
* Being 18 years of age or older.
* Knowing and understanding the Spanish language.
* Completing the informed consent.

Exclusion Criteria:

* The presence of any pathology in the family member that keeps the intervention from being carried out (such as psychosis, schizophrenia, intellectual disability, substance dependence, etc.) will be an exclusion criterion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Record of critical family-patient incidents | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  Number of Binge eating and vomiting episodes (purging) in the past 3 months, Number of serious arguments between patient and caregivers in the past 3 months, Number of days of self-injury in the past 3 months, Number of episodes of verbal/physical violence with caregivers in the past 3 months; Number of visits to psychiatric emergency department in the past 3 months, Number of unscheduled therapy sessions held in the past 3 months (face-to-face, phone calls, etc.).
Burden Assessment Scale (BAS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  It is a 19-item scale that assesses the caregiver's objective and subjective burden due to the illness of his/her loved one within the past six months using a 4-point Likert scale ranging from 1 (nothing) to 4 (a lot). Total scores indicate that higher values mean stronger burden. The scale shows adequate validity and reliability (Cronbach's alpha ranges from .89 to .91) (Reinhard, Gubman, Horwitz & Minsky, 1994).

SECONDARY OUTCOMES:
The Eating Disorder Symptom Impact Scale (EDSIS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  It is a 24-item scale to assess eating disorder-specific caregiving experiences using a 5-point Likert-type scale from 0 (Never) to 4 (Nearly Always). The internal consistency is good, with Cronbach's alpha coefficients mostly above .70.
Family Assessment Device - Global Functioning Scale | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  It is a 60-item self-report about family functioning in terms of problem-solving, communication, roles, affective responsiveness, affective involvement, behavior control, and general functioning. Items are rated on a 4-point Likert scale ranging from 1 (Completely Agree) to 4 (Strongly Disagree). The internal consistency is good (Cronbach's alphas between .72 and .83) for the subscales, with a Cronbach's alpha of .92 for general functioning.
Mastery and Empowerment Scale (MES) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  It is a 34-item scale divided into three domains: family, service system, and involvement in community. Items are rated on a 5-point Likert scale ranging from 1 (Completely False) to 5 (Completely True). Different studies have demonstrated that the psychometric properties of the FES are robust in both the original and translated versions (Koren et al., 1992; Singhet al., 1995; Itzhaky & Schwartz, 2001; Vuorenmaa et al., 2014).
Multicultural Quality of Life Index (MQLI) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  The Multicultural Quality of Life Index is a culture-informed and self-rated instrument. Its 10 items cover key aspects of the concept, from physical well-being to spiritual fulfilment. Regarding its applicability, mean completion time was less than 3 minutes, and 96% of raters found it easy to use. Test-retest reliability was high (r=0.87). A Cronbach's alpha of 0.92 documented its internal consistency, and a factor analysis revealed a strong structure.
The Multidimensional Existential Meaning Scale (MEMS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  It is a 15-item scale that assesses existential meaning through three dimensions: comprehension, purpose, and mattering. Items are rated on a 7-point Likert scale ranging from 1 (Very strongly disagree) to 7 (Very strongly agree). The three MEMS subscales showed adequate internal consistency: Comprehension (ω- = 91), Purpose (ω- = 92), and Mattering (ω- = 86).
Depression, Anxiety and Stress Scale (DASS-21). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  It is a 21-item scale in its short version that measures clinical symptoms such as depression, anxiety, and stress. Items are rated on a 4-point Likert scale ranging from 0 (It did not happen to me) to 3 (It happened to me a lot or most of the time). It shows excellent internal consistency: depression (α = .94), anxiety (α = .87), and stress (α= .91).
Difficulties in Emotion Regulation Scale (DERS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  In its adaptation, the authors reduced the items from 36 to 28, and they considered 5 scales instead 6. The subscales are: lack of emotional control, vital interference, lack of emotional attention, emotional confusion, and emotional rejection. Items are rated on a Likert-type scale ranging from 1 to 5 (1 = "Almost never" and 5 "Almost always"). Higher scores indicate greater difficulties with emotional regulation. Psychometric properties were adequate, with very good internal consistency (α = .93) and good test-retest reliability (pl = .74, p < .001).

OTHER OUTCOMES:
Opinion of treatment scale | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  This scale was designed and developed by members of the research team and constructed from an adaptation of another opinion and expectations questionnaire. The constructs this scale assesses are: opinion, acceptance and satisfaction with the skills training program, and the changes in the participants after the completion of each module. The questions refer to the rationale for the intervention, recommending the program, satisfaction with the program, usefulness, and expectations of the skills training. The items are rated on a Likert-type scale ranging from 0 "Not at all" to 10 "Very much".
The Eating Attitudes Test-26 (EAT-26) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  This scale is used to evaluate the patients. It is a 26-item self-report to assess attitudes toward eating. Items are rated on a 6-point Likert scale ranging from 1 (Never) to 6 (Always). The reliability analysis indicates good internal consistency Doninger, Enders, & Burnett, 2005; Garner etal., 1982; Jorquera, et al, 2006; Nunes, Camey, Olinto, &Mari, 2005; Pereira et al., 2008).
Patient Health Questionnaire (PHQ-9) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  This scale is used to evaluate the patients. It assesses each of the 9-DSM-IV criteria for depression in 9 items. Items are rated on a 4-point Likert scale ranging from 0 (Not at all) to 3 (Nearly Every Day).
Overall Anxiety Severity and Impairment Scale (OASIS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  This scale is used to evaluate the patients. It is a 5-item scale that assesses the severity and frequency of anxiety symptoms, behavioral avoidance, and the functional impairment related to anxiety. Items are rated on a 4-point Likert scale ranging from 0 to 4. The scale shows good psychometric properties such as test-retest reliability and internal consistency (α =.80).
Validating and Invalidating Responses Scale (VIRS). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  This scale is used to evaluate the patients. It is a 16-item scale that assesses the levels of perceived validation and invalidation of caregivers' responses, divided into validating and invalidating responses. Items are rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Almost Always). Higher scores signify greater perceived validation or invalidation of the responses of the caregiver being assessed.
Lum Emotional Availability of Parents (LEAP). | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 12-month follow-up
  This scale is used to evaluate the patients. It is a 15-item questionnaire that assesses the emotional availability of mothers and fathers as perceived by the person assessing their relatives. Items are rated on a 6-point Likert scale ranging from 1 (Never) to 6 (Always). The psychometric properties are very good, such that, in a clinical sample, excellent internal consistency is observed (for the mother α = .92, and for the father α = .93). In addition, it has adequate test-retest reliability for the mother's form (r = .92) and the father's form (r = .85).

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Fernández-Felipe, Study Chair — Universitat Jaume I de Castellón; Joaquín García-Alandete, Dr, Study Chair — University of Valencia; Sandra Pérez, Dr, Study Chair — University of Valencia; Sara Fonseca-Baeza, Study Chair — University of Valencia; Azucena García Palacios, Dr, Study Chair — Universitat Jaume I de Castellón; Rosa Baños, Dr., Study Chair — University of Valencia; Cristina Botella, Dr, Study Chair — Universitat Jaume I de Castellón
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after de-identification. Supporting Information:
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available immediately after publication
Access Criteria: The data will be available to anyone who wishes to access them

REFERENCES:
- [Result] Hoffman PD, Fruzzetti AE, Buteau E, Neiditch ER, Penney D, Bruce ML, Hellman F, Struening E. Family connections: a program for relatives of persons with borderline personality disorder. Fam Process. 2005 Jun;44(2):217-25. doi: 10.1111/j.1545-5300.2005.00055.x. PMID 16013747
- [Result] Dimitropoulos G, Landers A, Freeman V, Novick J, Schmidt U, Olmsted M. A feasibility study comparing a web-based intervention to a workshop intervention for caregivers of adults with eating disorders. Eur Eat Disord Rev. 2019 Nov;27(6):641-654. doi: 10.1002/erv.2678. Epub 2019 May 7. PMID 31063264
- [Result] Gisladottir M, Treasure J, Svavarsdottir EK. Effectiveness of therapeutic conversation intervention among caregivers of people with eating disorders: quasi-experimental design. J Clin Nurs. 2017 Mar;26(5-6):735-750. doi: 10.1111/jocn.13412. Epub 2016 Dec 7. PMID 27239974
- [Result] Grover M, Williams C, Eisler I, Fairbairn P, McCloskey C, Smith G, Treasure J, Schmidt U. An off-line pilot evaluation of a web-based systemic cognitive-behavioral intervention for carers of people with anorexia nervosa. Int J Eat Disord. 2011 Dec;44(8):708-15. doi: 10.1002/eat.20871. Epub 2010 Nov 15. PMID 22072408
- [Result] Hoffman PD, Fruzzetti AE. Advances in interventions for families with a relative with a personality disorder diagnosis. Curr Psychiatry Rep. 2007 Feb;9(1):68-73. doi: 10.1007/s11920-007-0012-z. PMID 17257517
- [Result] Flynn D, Kells M, Joyce M, Corcoran P, Herley S, Suarez C, Cotter P, Hurley J, Weihrauch M, Groeger J. Family Connections versus optimised treatment-as-usual for family members of individuals with borderline personality disorder: non-randomised controlled study. Borderline Personal Disord Emot Dysregul. 2017 Aug 30;4:18. doi: 10.1186/s40479-017-0069-1. eCollection 2017. PMID 28861273
- [Derived] Guillen V, Arnal A, Perez S, Garcia-Alandete J, Fernandez-Felipe I, Grau A, Botella C, Marco JH. Family connections in the treatment of relatives of people with eating disorders and personality disorders: study protocol of a randomized control trial. BMC Psychol. 2023 Mar 30;11(1):88. doi: 10.1186/s40359-023-01138-x. PMID 36998024